CLINICAL TRIAL: NCT01979952
Title: A Six Month Double Blind Randomized Placebo Controlled Trial Followed by Each Arm Being Converted to Oral Nintedanib 150 mg Twice Daily Comparing the Effect on High Resolution Computerized Tomography Quantitative Lung Fibrosis Score, Lung Function, Six Minute Walk Test Distance and St. George's Respiratory Questionnaire After Six Months of Treatment in Patients With Idiopathic Pulmonary Fibrosis With Continued Evaluations Over a Period of up to Eighteen Months
Brief Title: Nintedanib Twice Daily vs Placebo in Patients Diagnosed With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.187
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

ARMS (2):
- Nintedanib (Experimental): 150 mg twice daily
  Interventions: Drug: Nintedanib
- Placebo (Placebo Comparator): twice daily dosing
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Matching Placebo — twice daily dosing
  Arms: Placebo
Drug: Nintedanib — gelating capsule
  Arms: Nintedanib

SUMMARY:
This is an 6 month multi-centre, prospective, randomized, placebo controlled, double blind clinical trial followed by conversion of each arm to active nintedanib for an additional 6 months comparing the effect of nintedanib 150mg bis in die (BID twice daily) on the progression of IPF measured by using High Resolution Computerized Tomography(HRCT), lung function, functional component (6MWT), biomarkers, and PRO component (PROs) with continued treatment and assessments for up to 18 months.

ELIGIBILITY:
Inclusion criteria:

1. Written Informed Consent consistent with International Conference on Harmonisation Good Clinical Practice (ICH-GCP) and local laws signed prior to entry into the study
2. Patient aged >= 40 years at Visit 1.
3. IPF diagnosed, according to the 2011 American Thoracic Society (ATS) / European Respiratory Society (ERS) / Japanese Respiratory Society(JRS)/ Latin American Thoracic Association (ALAT)/ Latin American Thoracic Association/ Idiopathic Pulmonary Fibrosis (IPF) guidelines for diagnosis and management, within 5 years and reaffirmed applying 2011 Guidelines (P11-07084) if diagnosed >2 years and up to 5 year from Visit 1,. Diagnosis must be confirmed by chest High Resolution Computerized Tomography (HRCT) taken within 24 months of Visit 1. All HRCT results reported to be possible or inconsistent usual interstitial pneumonia (UIP) must have confirmatory pathology.
4. Carbon monoxide Diffusing capacity or Transfer factor of the lung for carbon monoxide (DLCO) (corrected for Hb): 30%-79% predicted of normal
5. Forced Vital Capacity (FVC) >= 50% predicted of normal at Visit 1 and Visit 2

Exclusion criteria:

1. AST, ALT > 1.5 fold ULN
2. Bilirubin > 1.5 fold ULN
3. Bleeding risk:

   1. Patients who require fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, dabigatran, heparin, hirudin), or high dose antiplatelet therapy. Exceptions: prophylactic low dose heparin or heparin flush as needed for maintenance of an indwelling intravenous device (e.g. enoxaparin 4000 IU s.c. per day) and prophylactic use of antiplatelet therapy (e.g. acetyl salicylic acid up to 325 mg/d, or clopidogrel at 75 mg/d, or equivalent doses of other antiplatelet therapy)
   2. History of hemorrhagic Central Nervous System (CNS) event within 12 months
   3. Any of the following within 3 months:

      * Haemoptysis or haematuria.
      * Active gastro-intestinal bleeding or ulcers.
      * Major injury or surgery.
   4. Coagulation parameters: International normalised ratio (INR) > 2, prothrombin time (PT) and partial thromboplastin time (PTT) > 150% of institutional ULN.
4. Planned major surgery within the next 3 months, including lung transplantation, major abdominal or major intestinal surgery.
5. Thrombotic risk

   1. Known inherited predisposition to thrombosis.
   2. History of thrombotic event (including stroke and transient ischemic attacks) within 12 months
6. Current or planned usage of any investigational drug during the course of this trial
7. Previous treatment with nintedanib within a clinical trial in the previous 3 months and discontinuation of nintedanib study treatment due to an adverse event
8. Known hypersensitivity to the trial drug or its component
9. A disease or condition which in the opinion of investigator may put the patient at risk because of participation in this trial or limit the patient's ability to participate in this trial. Patients will be excluded if they require greater than 12L/min oxygen, are not ambulatory or require use of a walker or cane during the 6 Minute Titration Walk Test. Patients who cannot complete the 6 Minute Titration Walk Test are excluded from participation.
10. Alcohol or drug abuse which in the opinion of the investigator would interfere with trial participation.
11. Pregnant women or women who are breast feeding or of child bearing potential not using two effective methods of birth control (one barrier and one highly effective non-barrier) for at least 1 month prior to trial and/or not committing to using it until 3 months after end of treatment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2016-10-27 (Actual); Study Completion 2016-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (25):
- United States (11):
  - Western CT Medical Group, P.C., Danbury, Connecticut
  - Clinical Research Center Sarasota Memorial Hosptial, Sarasota, Florida
  - Chest Medicine Clinical Services, Skokie, Illinois
  - Baptist Health Lexington, Lexington, Kentucky
  - Minnesota Lung Research, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Winthrop University Hospital, Mineola, New York
  - ID Clinical Research, LTD, Toledo, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Lowcountry Lung and Crit Care, Charleston, South Carolina
  - Annette C & Harold C Simmons Transplant Institute, Dallas, Texas
- Canada (7):
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Concordia Hospital, Winnipeg, Manitoba
  - QEII Health Sciences Centre (Dalhousie University), Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - CHUS Fleurimont, Sherbrooke, Quebec
- Turkey (Türkiye) (7):
  - Cukurova Universitesi Tip Fakultesi Gog. Hast. Anabilim Dali, Adana
  - Ankara Universitesi Tip Fakultesi, Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Yedikule Gog. Hst. EAH, Istanbul
  - Sureyyapasa Gogus Hast. ve Gogus Cer. Egit. ve Aras. Has., Istanbul
  - Ege Universitesi T.F., Izmir
  - Dr.Suat Seren EAH, Izmir

REFERENCES:
- [Derived] Glaspole I, Bonella F, Bargagli E, Glassberg MK, Caro F, Stansen W, Quaresma M, Orsatti L, Bendstrup E. Efficacy and safety of nintedanib in patients with idiopathic pulmonary fibrosis who are elderly or have comorbidities. Respir Res. 2021 Apr 26;22(1):125. doi: 10.1186/s12931-021-01695-y. PMID 33902584

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized to receive nintedanib or placebo in 1:1 ratio. After Global Amendment 1, study design was changed to exploratory, and duration of double blind, placebo-controlled part of study was reduced from 12 months to 6 months, followed by conversion of all patients to open-label nintedanib treatment for a duration of up to 18 months.
Groups:
- Nintedanib: Patients received oral administration of 150 milligram (mg) soft gelatin capsules of nintedanib (Ofev ®) twice daily for up to 18 months.
- Placebo: Patients receive oral administration of matching placebo of 150 mg nintedanib twice daily for a period of at least 6 months after randomization
Period: Overall Study
Arm/Group | Nintedanib | Placebo
Started | 56 | 57
Completed | 48 | 51
Not Completed | 8 | 6
Not completed — Adverse Event | 4 | 5
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other than specified above | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) consisted of patients who were randomized to a treatment group and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib | Placebo | Total
Number analyzed (Participants) | 56 | 57 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.8 (7.6) | 66.2 (9.4) | 67.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 20 | 31
  Male | 45 | 37 | 82

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in High Resolution Computerized Tomography (HRCT) Quantitative Lung Fibrosis (QLF) Score at 6 Months
Description: Relative change from baseline in HRCT QLF score at 6 months was calculated as the difference of the QLF score at month 6 minus the QLF score at baseline divided by the baseline QLF score. The QLF score itself ranges from 0 to 100%, where greater values represent a greater amount of lung fibrosis and are considered a worse health status. Hence smaller relative changes from baseline (i.e., ratios) were considered favorable. HCRT assessment obtained during screening visit was considered as baseline.
Time Frame: Baseline and 6 Months
Population: Observed Cases (6 months) (OC6): The OC6 consisted of all patients in the TS (all patients who were randomized to a treatment group and received at least 1 dose of study drug) with observed data for the primary endpoint (relative change from baseline in HRCT QLF score at 6 months).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 42 | 45
percent change | 11.407 (4.4819) | 14.583 (4.3297)
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; Analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline HRCT QLF score as covariate; Test type: Superiority or Other; ANCOVA; As per the Clinical Trial Protocol, this is an exploratory trial hence p-values were not calculated; Adjusted mean difference = 3.176, 95% CI 2-sided [-9.227 to 15.579], Standard Error of Mean 6.2370

2. Secondary Outcome: Effect of Six Month Delayed Treatment Onset: Relative Change From Baseline in HRCT QLF Score at 12 Months
Description: Relative change from baseline in HRCT QLF score at 12 months was calculated as the ratio of the QLF score at 12 months to baseline. Greater values of the QLF score represented a worse health status and hence smaller relative changes from baseline (i.e., ratios) were considered favorable.
  HCRT assessment obtained during screening visit was considered as baseline. Note that due to the change in study design, patients randomized to the placebo group were treated with nintedanib after completion of the first 6-month treatment period. Therefore, this new endpoint was defined to address the effect of a 6-month delayed onset of nintedanib treatment.
Time Frame: Baseline and 12 Months
Population: Observed Cases (12 months) (OC12): The OC12 consisted of all patients in OC6 with observed QLF data at 12 months.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 30 | 31
percent change | 13.103 (4.5454) | 15.622 (4.4714)
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; Analysis of covariance (ANCOVA) model with treatment as fixed effect and baseline HRCT QLF score as covariate; Test type: Superiority or Other; ANCOVA; As per the Clinical Trial Protocol, this is an exploratory trial hence p-values were not calculated; Adjusted mean difference = 2.519, 95% CI 2-sided [-10.258 to 15.296], Standard Error of Mean 6.3829

3. Secondary Outcome: Absolute Change in Forced Vital Capacity (FVC) From Baseline at 6 Months
Description: Absolute change in Forced Vital Capacity (FVC) from baseline at 6 months is presented.
Time Frame: Baseline and 6 Months
Population: Treated Set (TS) (Only patients with observed cases (OC) values were analysed)
Measure: Least Squares Mean (Standard Error); unit: milliliter (mL)
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 54 | 54
milliliter (mL) | -14.18 (31.050) | -83.18 (28.067)
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; Mixed Model for Repeated Measures (MMRM) model with fixed effects for treatment, visit, gender, age, height, treatment-by-visit, baseline FVC, baseline FVC-by-visit and random effect for patient. Within-patient errors are modelled by unstructured covariance matrix; Test type: Superiority or Other; Mixed Models Analysis; As per the Clinical Trial Protocol, this is an exploratory trial hence p-values were not calculated; Adjusted mean difference = 69.00, 95% CI 2-sided [-8.74 to 146.75], Standard Error of Mean 39.182

4. Secondary Outcome: Relative Change in FVC From Baseline at 6 Months
Description: Relative change in FVC from baseline at 6 months is presented.
Time Frame: Baseline and 6 Months
Population: TS (Only patients with observed cases (OC) values were analysed)
Measure: Least Squares Mean (Standard Error); unit: percentage of change
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 54 | 54
percentage of change | -0.67 (1.05) | -3.02 (0.95)
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; MMRM model with fixed effects for treatment, visit, gender, age, height, treatment-by-visit, baseline FVC, baseline FVC-by-visit and random effect for patient. Within-patient errors are modelled by unstructured covariance matrix; Test type: Superiority or Other; Mixed Models Analysis; As per the Clinical Trial Protocol, this is an exploratory trial hence p-values were not calculated; Adjusted mean difference = 2.36, 95% CI 2-sided [-0.29 to 5.00]

5. Secondary Outcome: Categorical Change in FVC From Baseline at 6 Months
Description: Percentage of participants reporting categorical change in FVC from baseline at 6 months are presented.
Time Frame: Baseline and 6 Months
Population: TS (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: Percentage of participants
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 46 | 46
Percentage of participants
  Decrease >10% or 200 mL | 6.5 | 23.9
  Change within ≤10% AND ≤200 mL | 76.1 | 71.7
  Increase >10% or 200 mL | 17.4 | 4.3

6. Secondary Outcome: St. George's Respiratory Questionnaire (SGRQ) Total Score Change From Baseline at 6 Months
Description: SGRQ total score change from baseline at 6 months is presented. SGRQ is a health-related quality of life questionnaire divided into 3 components : symptoms, activity and impact.
  The total score (summed weights) can range from 0 to 100 with a lower score denoting a better health status.
  Means provided are the adjusted means based on all analyzed patients in the model (not only patients with a baseline and measurement at month 6).
Time Frame: Baseline and 6 Months
Population: TS (Only patients with observed cases (OC) values were analysed)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 55 | 53
Units on a scale | -2.24 (1.682) | -2.19 (1.699)
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; MMRM model included treatment, visit, baseline value, treatment-by-visit and baseline-by-visit as fixed effects and patient as random effect. Unstructured covariance was assumed for within patient variation; Test type: Superiority or Other; Mixed Models Analysis; Adjusted mean difference = -0.05, 95% CI 2-sided [-4.89 to 4.79], Standard Error of Mean 2.434

7. Secondary Outcome: 6MWT Total Distance Walked Change From Baseline at 6 Months
Description: Change in total distance covered in 6-minute walk test (6MWT) from baseline at 6 month is presented.
  The 6-Minutes Walk Test (6-MWT) was conducted according to the American Thoracic Society (ATS) Criteria.
Time Frame: Baseline and 6 Months
Population: TS (Only patients with observed cases (OC) values were analysed)
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 55 | 52
meters | 4.93 (11.415) | -13.00 (11.476)
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Adjusted mean difference = 17.94, 95% CI 2-sided [-14.21 to 50.09], Standard Error of Mean 16.190

8. Secondary Outcome: University of California San Diego Shortness of Breath Questionnaire (UCSD-SOBQ) Change From Baseline at 6 Months
Description: University of California San Diego Shortness of Breath Questionnaire (UCSD-SOBQ) change from baseline at 6 months is presented. Shortness of Breath Questionnaire measures the shortness of breath. It comprises of 24 items. Each item is scored on a scale between 0-5 where 5 represents maximal breathlessness. The responses to all items are summed up to provide the overall score that can range from 0 (best outcome) to 120 (worst outcome).
  Means presented are the adjusted means and are based on all analyzed patients in the model (not only patients with a baseline and measurement at month 6).
Time Frame: Baseline and 6 Months
Population: TS (Only patients with observed cases (OC) values were analysed)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 53 | 50
Units on a scale | 3.42 (2.156) | -1.46 (2.192)
Statistical Analysis 1: Comparison: Nintedanib vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Adjusted mean difference = 4.89, 95% CI 2-sided [-1.47 to 11.25]

9. Secondary Outcome: All-cause Mortality at 6 Months
Description: Percentage of subjects died from all causes between 0 to 6 months are presented.
Time Frame: 6 Months
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 56 | 57
Percentage of participants | 0.0 | 5.3

10. Secondary Outcome: Respiratory Hospitalizations at 6 Months
Description: Percentage of subjects hospitalized due to respiratory problems between 0 to 6 months are presented.
Time Frame: 6 Months
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 56 | 57
Percentage of participants | 0.0 | 7.0

11. Secondary Outcome: Respiratory Mortality at 6 Months
Description: Percentage of subjects who died due to respiratory cause between 0 to 6 months are presented.
Time Frame: 6 Months
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 56 | 57
Percentage of participants | 0.0 | 3.5

12. Secondary Outcome: Acute Idiopathic Pulmonary Fibrosis (IPF) Exacerbations at 6 Months
Description: Percentage of subjects experienced first acute IPF exacerbations (based on Investigator reported adverse events) between 0 to 6 months are presented.
Time Frame: 6 Months
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | Nintedanib | Placebo
Number analyzed (Participants) | 56 | 57
Percentage of participants | 1.8 | 1.8

ADVERSE EVENTS:
Time Frame: From first drug administration till 28 days after end of treatment; up to 19 months
Description: Treated Set
Arm/Group | Nintedanib | Placebo
Serious Adverse Events (participants affected / at risk) | 11/56 | 14/57
Other Adverse Events (participants affected / at risk) | 54/56 | 51/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=56) | Placebo (N=57)
Cardiogenic shock (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lyme disease (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=56) | Placebo (N=57)
Eosinophilia (Blood and lymphatic system disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 5
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 43 | 40
Flatulence (Gastrointestinal disorders) | 0 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 16 | 20
Vomiting (Gastrointestinal disorders) | 10 | 9
Asthenia (General disorders) | 0 | 3
Fatigue (General disorders) | 11 | 9
Bronchitis (Infections and infestations) | 4 | 7
Influenza (Infections and infestations) | 8 | 6
Lower respiratory tract infection (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 5 | 9
Respiratory tract infection (Infections and infestations) | 4 | 3
Sinusitis (Infections and infestations) | 3 | 3
Tooth abscess (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 7
Urinary tract infection (Infections and infestations) | 3 | 5
Fall (Injury, poisoning and procedural complications) | 1 | 4
Alanine aminotransferase increased (Investigations) | 3 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 3
Eosinophil count increased (Investigations) | 4 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 3
International normalised ratio increased (Investigations) | 3 | 1
Prothrombin time prolonged (Investigations) | 3 | 1
Weight decreased (Investigations) | 13 | 4
Decreased appetite (Metabolism and nutrition disorders) | 12 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Dizziness (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 7 | 9
Depression (Psychiatric disorders) | 2 | 3
Nephrolithiasis (Renal and urinary disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 3 | 4

LIMITATIONS AND CAVEATS:
This study was an exploratory trial that was not statistically powered to demonstrate significant differences between treatment groups for the efficacy endpoints evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.